CLINICAL TRIAL: NCT00005308
Title: Anemia and Surgery: Indications For Transfusion
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 3011; R01HL041523 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2001-11

CONDITIONS: Blood Disease; Anemia
MeSH Terms: conditions — Hematologic Diseases; Anemia

SUMMARY:
To estimate the risk of death for patients with different pre- and post-operative hemoglobin levels who do not receive blood transfusions and to derive a multivariate model using clinical information available pre-operatively that would predict the risk of death post-operatively.

DETAILED DESCRIPTION:
BACKGROUND:

The AIDS epidemic has focused considerable attention on the risks associated with blood transfusions. Perhaps of more importance, hemolytic transfusion reactions and post-transfusion non-A non-B hepatitis continue to be significant concerns. However, guidelines for blood transfusions in the surgical patient vary considerably in the medical literature. Some recent texts stress the need to consider factors such as patient's age, surgical procedure, co-morbid illness, predicted blood loss, and cause of the anemia, as well as the hemoglobin level. Nonetheless, in practice many surgeons still adhere to the 10g/dl threshold for transfusion. The lack of consensus guidelines can probably be attributed to the dearth of studies exploring the indications for transfusion. The few studies which have examined this question are limited because they fail to analyze subsets of patients by age, co-morbid illness, or blood loss. The need to develop peri-operative transfusion guidelines based on multivariate analysis, therefore decreasing the frequency of unnecessary transfusions resulting from the common use of a hemoglobin threshold, is especially important in light of the hazards and costs associated with blood transfusions. Jehovah's Witnesses were chosen as the study population because they decline blood transfusion for religious reasons.

DESIGN NARRATIVE:

The retrospective case-control study explored the possible associations between peri-operative anemia and post-operative mortality status. Cases were defined as those who died within 30 days of the operative procedure and controls as all those who survived. There were approximately eight controls per case. Participating surgeons who operated on Jehovah's Witness patients within the preceeding five years provide a list of patients. Charts of patients were reviewed to determine if any died within 30 days of surgery. If the patient was discharged prior to 30 days postoperatively, then the National Death Index was used to assess the patient's status 30 days after surgery. The incidence of post-operative death, with 95 percent confidence levels, was calculated for strata of pre- and post-operative hemoglobin levels and operative blood loss. The death rate was calculated after stratifying the patients based on status with regard to co-morbid diseases or other possible risk factors.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-04; Study Completion 1995-03 (Actual)